CLINICAL TRIAL: NCT07105345
Title: Efficacy of Multi-Modal Cognitive Processing Therapy for PTSD: A Longitudinal, Multicenter, Single-Blind RCT on Symptoms, Sleep, Anxiety, Depression, Remission, and Posttraumatic Growth
Brief Title: Exploring Efficacy of Multi-Mode Cognitive Processing Therapy (CPT) for PTSD
Acronym: PTSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FEMH No.：114037-F; IRB FEMH No.：114037-F (Other: Far Eastern Memorial Hospital)
Record Dates: First submitted 2025-06-23; First posted 2025-08-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Cognitive Processing Therapy; Trauma-focused therapy; Sleep quality; Anxiety; RCT; Taiwan; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial with participants assigned to either CPT or TAU.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to group assignment to reduce bias in post-intervention evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Processing Therapy (CPT) (Experimental): Participants in this arm will receive 12 weekly individual sessions of Cognitive Processing Therapy (CPT), based on the Resick protocol. Each session will last 90 minutes and will be delivered by a trained therapist. The therapy integrates cognitive restructuring, trauma-related belief processing, and behavioral assignments.
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)
- Treatment as Usual (TAU) (Active Comparator): Participants in this group will receive routine outpatient psychiatric care as determined by their clinician, which may include medication, general supportive therapy, or psychoeducation, but will not include structured CPT sessions.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — Participants will receive 12 weekly 90-minute individual sessions of Cognitive Processing Therapy (CPT) following the Resick manual. The intervention includes cognitive restructuring, trauma-related belief processing, and structured behavioral assignments. Sessions are delivered by trained therapists.
  Other Names: MMCPT
  Arms: Cognitive Processing Therapy (CPT)
Other: Treatment as Usual (TAU) — Participants will receive routine outpatient psychiatric care as determined by clinicians. This may include medication, general supportive therapy, or psychoeducation, but will not include structured CPT sessions.
  Other Names: Standard psychiatric care
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study is a longitudinal, multicenter, single-blind, two-arm randomized controlled trial designed to evaluate the effectiveness of Multi-Modal Cognitive Processing Therapy (MMCPT) for individuals with posttraumatic stress disorder (PTSD). Participants will be randomly assigned to either the intervention group receiving MMCPT or a control group receiving treatment-as-usual (TAU). The intervention follows the standard CPT manual developed by Resick and consists of twelve weekly 90-minute individual sessions. The primary outcomes include PTSD symptom severity assessed by the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) and the PTSD Checklist for DSM-5 (PCL-5). Secondary outcomes include sleep quality (actigraphy, PSQI), anxiety (STAI), depression (HDRS-17), remission rate, and posttraumatic growth (PTGI). Assessments will occur at baseline, mid-treatment, post-treatment, and at 3-, 6-, 9-, and 12-month follow-ups.

DETAILED DESCRIPTION:
This clinical trial aims to construct and evaluate a multi-modal Cognitive Processing Therapy (MMCPT) model and examine its long-term effects on PTSD symptoms, sleep, anxiety, depression, remission, and posttraumatic growth. The study employs a longitudinal, multicenter, single-blind randomized controlled design with two parallel arms. Participants diagnosed with PTSD at psychiatric outpatient clinics will be randomized to either MMCPT or TAU. The MMCPT follows the CPT manual developed by Resick and includes twelve 90-minute weekly individual sessions delivered by fully trained therapists.

The primary outcomes are PTSD symptom severity measured by CAPS-5 and PCL-5. Secondary outcomes include sleep quality measured via actigraphy and the Pittsburgh Sleep Quality Index (PSQI), anxiety levels via the State-Trait Anxiety Inventory (STAI), depression severity via the Hamilton Depression Rating Scale (HDRS-17), remission rate via CAPS-5 and PCL-5, and posttraumatic growth via the Posttraumatic Growth Inventory (PTGI).

Assessments are scheduled at seven time points: pre-treatment, mid-treatment (after session 6), post-treatment (after session 12), and follow-up at 3, 6, 9, and 12 months. The study also includes training and supervision of therapists and evaluators, as well as rigorous monitoring of allocation concealment, treatment fidelity, dropout, medication use, blinding, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 65 years
* Diagnosed with PTSD according to DSM-5 criteria
* Score ≥ 33 on the PTSD Checklist for DSM-5 (PCL-5)
* Able to provide informed consent
* Stable psychiatric medication regimen (if any) for at least 4 weeks prior to enrollment

Exclusion Criteria:

* Diagnosed with schizophrenia, schizoaffective disorder, or bipolar I disorder
* Current substance dependence or abuse within the past 6 months
* Severe suicidal ideation or suicide attempt in the past 6 months
* Cognitive impairment or neurological disorder affecting participation
* Concurrent participation in other psychological treatment for PTSD

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptom severity (CAPS-5) | Baseline (Screening Visit, prior to randomization)
  PTSD symptom severity will be measured using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). The total score ranges from 0 to 80, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Change in PTSD symptoms (PCL-5) | Baseline, Week 6 ( Mid-treatment), Week 12 (Post-treatment), Month 3, Month 6, Month 9, and Month 12 follow-up
  Self-reported PTSD symptoms will be assessed using the PTSD Checklist for DSM-5 (PCL-5). The score ranges from 0 to 80; higher scores indicate more severe symptoms.
Sleep quality (PSQI score and actigraphy) | Baseline, Week 6 ( Mid-treatment), Week 12 (Post-treatment), Month 3, Month 6, Month 9, and Month 12 follow-up
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) and actigraphy monitoring. The PSQI score ranges from 0 to 21.
Anxiety symptoms (STAI) | Baseline, Week 6 ( Mid-treatment), Week 12 (Post-treatment), Month 3, Month 6, Month 9, and Month 12 follow-up
  Anxiety severity will be measured using the State-Trait Anxiety Inventory (STAI). Each subscale score ranges from 20 to 80.
Depression symptoms (HDRS-17) | Baseline, Week 6 ( Mid-treatment), Week 12 (Post-treatment), Month 3, Month 6, Month 9, and Month 12 follow-up
  Depression severity will be assessed using the 17-item Hamilton Depression Rating Scale (HDRS-17). The total score ranges from 0 to 52, with higher scores indicating more severe depression symptoms.
Posttraumatic growth (PTGI) | Baseline, Week 6 ( Mid-treatment), Week 12 (Post-treatment), Month 3, Month 6, Month 9, and Month 12 follow-up
  Posttraumatic growth will be assessed using the Posttraumatic Growth Inventory (PTGI). The total score ranges from 0 to 105, with higher scores indicating greater posttraumatic growth.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Banqiao District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Due to privacy and ethical considerations, no plan to share individual participant data (IPD) has been determined at this time. If data sharing is considered in the future, it will follow IRB approval and data use request procedures.